CLINICAL TRIAL: NCT03586804
Title: Comparison of Postural Sway Responses at Menstrual Cyclus in Women With and Without Dysmenorrheal Syndrome
Brief Title: Postural Sway at Menstrual Cyclus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Assoc Prof,PhD, Hacettepe University
Other Study IDs: TU-216
Record Dates: First submitted 2018-07-06; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Women's Health: Endometriosis
Keywords: menstrual; postural sway; dual task

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women without dysmenorrheal syndrome: women without dysmenorrheal syndrome
  Interventions: Other: dual task
- women with dysmenorrheal syndrome: women with dysmenorrheal syndrome
  Interventions: Other: dual task

INTERVENTIONS:
Other: dual task — mental and motor tasks will be performed while standing. Motor task: holding mini blocks Mental task: Counting the numbers from 200 to 1

SUMMARY:
The study was planned with the aim of comparison of postural sway responses at menstrual cycles in women with and without the dysmenorrheal syndrome.

Women will stand on a postural sway evaluation system on the first day of the menstrual cycles and a well-being day which they will select. Every participant will be evaluated same tool. They will be assessed for three times at every session: 1st evaluation will be performed at the normal standing position. 2nd evaluation will be performed at the normal standing position while individuals saying the numbers from 200 to 1. 3rd evaluation will be performed at the normal standing position while individuals holding the mini blocks on their hands.

DETAILED DESCRIPTION:
The study was planned with the aim of comparison of postural sway responses at menstrual cycles in women with and without the dysmenorrheal syndrome.

Women will stand on a postural sway evaluation system on the first day of the menstrual cycles and a well-being day which they will select. Every participant will be evaluated with the same tool. They will be assessed for three times at every session: 1st evaluation will be performed at the normal standing position. 2nd evaluation will be performed at the normal standing position while individuals saying the numbers from 200 to 1. 3rd evaluation will be performed at the normal standing position while individuals holding the mini blocks on their hands.

Results will be compared for menstrual cycles and well-being day in women with and without pain at menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Have dysmenorrheal syndrome
* Have menstrual cycle without pain

Exclusion Criteria:

* Have another health problem (systemic, neurologic, orthopedic or psychiatric)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with and without pain at menstrual cycles
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of Postural sway score | First evaluation: at first minute. Second evauation: Change baseline postural sway score at 15th minutes. Third evaluation: Change baseline postural sway score at 30th minutes.
  Postural sway is a swing of the body while a person is standing in upright position.

IPD SHARING:
Plan to Share IPD: Undecided